CLINICAL TRIAL: NCT03947151
Title: Efficacy and Tolerance of an Ovarian Stimulation Protocol Combining FSH and Degarelix Acetate in Female Candidates for Fertility Preservation Before Chemotherapy for Breast Cancer
Brief Title: Efficacy and Tolerance of an Ovarian Stimulation Protocol Combining Follicle Stimulating Hormone (FSH) and Degarelix Acetate in Female Candidates for Fertility Preservation Before Chemotherapy for Breast Cancer
Acronym: DEGASTIM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: P170407J; 2018-000049-38 (EudraCT Number)
Record Dates: First submitted 2019-01-17; First posted 2019-05-13 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Invasive Ductal Breast Carcinoma
Keywords: Fertility preservation; Controlled ovarian stimulation; Oocyte vitrification; GnRH antagonist protocol
MeSH Terms: conditions — Carcinoma, Ductal, Breast | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- one arm (Other): one arm
  Interventions: Drug: Degarelix injection(s)

INTERVENTIONS:
Drug: Degarelix injection(s) — 1 or 2 degarelix injection(s)
  Other Names: Firmagon®

SUMMARY:
The present investigation aims to evaluate the efficacy of an innovative protocol of controlled ovarian stimulation for breast cancer patients, who are candidates for fertility preservation.

Currently, vitrification of oocytes and/or embryos after controlled ovarian stimulation is the most established method for female fertility preservation. However, this stimulation induces an increase in serum estrogen levels, which is theoretically problematic in case of hormone-sensitive tumors such as breast cancer. The majority of oncology teams accept, in very specific situations (particularly when the tumor has been surgically removed), this ovarian stimulation, because the expected benefits of fertility preservation far outweigh the risks. However, everyone agrees that it would be more comfortable to be able to offer vitrification of oocytes and/or embryos using ovarian stimulation without increasing estrogen levels.

In this research, investigators will evaluate the efficacy of degarelix (Firmagon®), currently indicated for the treatment of prostate cancer, as an innovative ovarian stimulation procedure. Administered at the beginning of ovarian stimulation, they believe it should maintain serum estradiol levels at physiological values at the end of stimulation.

DETAILED DESCRIPTION:
Recent improvements in freezing techniques have led to the development of fertility preservation techniques for young women diagnosed with cancer. Currently, vitrification of oocytes or embryos after controlled ovarian stimulation (COS) represents the only established method. This COS is based on the daily administration of exogenous Follicle Stimulating Hormone (FSH) and an ovulation blockage using Gonadotropin Releasing Hormone (GnRH) antagonists (0.25 mg/d) initiated after approximately 6 days of stimulation and continued until ovulation is triggered.

In addition to requiring 15 days, COS induces supraphysiological hyperestradiolaemia (5-10 times normal) which can be problematic in case of hormone-sensitive tumors such as breast cancer. The majority of oncology teams accept, in very specific situations (particularly when the tumor has been surgically removed), this ovarian stimulation, because the expected benefits of fertility preservation far outweigh the risks. However, everyone agrees that it would be more comfortable to be able to offer vitrification of oocytes and/or embryos using ovarian stimulation without increasing estrogen levels.

Therefore, the limitation of serum estradiol concentrations during stimulation represents an important issue. To this end, stimulation protocols combining aromatase inhibitors have been proposed. Inhibition of the P450 aromatase enzyme in the granulosa cells of stimulated follicles prevents the conversion of androgens to estrogens. However, the teratogenic risk of these molecules, although discussed, limits their use in the indication of COS. Recently, a new "natos" protocol was proposed to stimulate the ovaries while maintaining physiological estradiolaemia, without using aromatase inhibitors. Thus, the administration of high doses of Gonadotropin Releasing Hormone (GnRH) antagonists (3 to 6 injections of 0.25 mg/day) from the beginning of COS, would allow a strong Luteinizing Hormone (LH) deprivation, thus limiting the production of androgens according to the 2 cells - 2 gonadotropins theory. In the absence of a precursor, estradiolemia remains at physiological ranges during the total duration of COS. However, the relative heaviness of a protocol combining up to 8 daily injections limits its use in young women who are candidates for fertility preservation.

Investigators therefore propose to evaluate the efficacy and tolerance of a new natos-like COS protocol based on the administration of a long-acting GnRH antagonist, degarelix. This drug is currently off-label for women.

The expected duration of the research is 14 months and participation will be 2 months.

After signature of the consent, during the first visit (oncofertility counseling), the the research (consultations and examinations) will be carried out within the Antoine Béclère hospital. All visits and examinations performed are part of routine care, except for the injection(s) of degarelix which belongs to the research.

Inclusion visit During the oncofertility consultation, the physician will make sure that the patient can be included in the research. Once the consent has been signed, the doctor will schedule the following visits based on the biological results obtained as part of the usual care.

Research follow-up visits

Stimulation: between the day of oncofertility counseling and the following 7 days, the doctor will check that patients are in the early follicular phase of the cycle, Degarelix injection: 1 injection, under the skin (possibly renewable after 5-7 days if the serum LH is ≥2 IU / L and / or the estradiol is ≥400 pg / mL), Concomitant initiation of ovarian stimulation by administration of recombinant FSH - Follitropin alfa (usual care). The injections will be given by the patient or a nurse at home, between 7pm and 10pm.

Stimulation follow-up visit #1 :

After 5 days of ovarian stimulation, transvaginal pelvic ultrasound (counting of ovarian follicles and measurement of their diameters) and blood sampling for serum hormone assays (estradiol, LH, progesterone) will be performed as part of the usual care.

Stimulation follow-up visits #2 and #3 Visits #2 and #3: transvaginal pelvic ultrasound (counting of ovarian follicles and measurement of their diameters) and a blood test for serum hormone assays (estradiol, LH, progesterone) will be required to monitor the response to stimulation, as part of routine care.

Visits are repeated until 4 follicles 16 to 20 mm in diameter are obtained, which is the criterion for ovulation trigger using 1 injection of Human Chorionic Gonadotropin (hCG) (Ovitrelle 250 mcg, SC) (usual care). Thus visits #2 and #3 are systematic. One or two additional visits with the same examinations may sometimes be necessary if the trigger criteria are not met.

Thirty-six hours after Human Chorionic Gonadotropin (hCG) , oocyte retrieval will be performed.

Visit on the day of the oocyte retrieval:

Patients will have a venous blood sample for serum hormone assays (estradiol, LH, progesterone) as part of the usual care.

Oocyte collection will be scheduled, and those which are mature will then be frozen (by vitrification) or fertilized in vitro in case of embryo freezing.

Visit following egg retrieval:

A blood test for serum hormone assays (estradiol, LH, progesterone) will be performed 3-4 days after oocyte retrieval.

End of research visit Participants will be contacted by phone 2 months after the injection of degarelix (Firmagon®) to make sure they are fine.

ELIGIBILITY:
Inclusion Criteria:

* Patients with invasive ductal carcinoma breast cancer, whatever the hormonal receptor expression profile
* Age : 18 - 40 years
* Presence of 2 ovaries
* Antral follicular count between 12 and 30 on both ovaries and/or recent measurement of serum anti-Müllerian hormone between 1.5 and 4 ng / mL (between Day-25 and Day0)
* Indication of chemotherapy
* Indication of preservation of fertility according to an oocyte vitrification technique after controlled ovarian stimulation (COS)
* Patient in the early follicular phase of the cycle at the start of the controlled ovarian stimulation (COS) (absence of follicle> 10 mm in ultrasound and estradiolemia <50 pg / mL)
* Oncology team agreement for the controlled ovarian stimulation (COS)
* Social insured patient
* Patient who gave her consent to participate by signing the consent of the study

Exclusion Criteria:

* Patient in late follicular phase or luteal phase
* Known hypersensitivity to one of the constituents of Firmagon®

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2019-11-28 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Number of follicles 16 to 20 mm in diameter obtained with estradiolemia <500 pg /mL | Day of ovulation trigger
  Success of the procedure if at least 4 follicles 16 to 20 mm in diameter are obtained on the day of ovulation trigger (36 hours before oocyte collection) with estradiolemia <500 pg / mL

SECONDARY OUTCOMES:
Serum estradiol levels | Day of ovulation trigger
Percentage of women with hyperestradiolemia | from the beginning of the controlled ovarian stimulation until Month 2
  Percentage of women with hyperestradiolemia during controlled ovarian stimulation (COS)
Duration of the increase in serum estradiol levels | from the beginning of the controlled ovarian stimulation until Month 2
Number of oocytes collected | through oocyte collection, an average of Day 20
  Outcome of ovarian stimulation evaluated by the number of oocytes collected, and the number of mature oocytes vitrified
Number of mature oocytes vitrified | through oocyte collection, an average of Day 20
  Outcome of ovarian stimulation evaluated by the number of oocytes collected, and the number of mature oocytes vitrified
Nature of serious side effects | 2 months
  Description : Serious side effects associated with treatment with degarelix (MedDRA coding)

CONTACTS AND LOCATIONS:
Overall Officials: Michaël GRYNBERG, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Antoine Béclère, Clamart, France